CLINICAL TRIAL: NCT05411016
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose or Multiple Ascending Dose Study of KK4277 in Healthy Volunteers, Patient With Systemic Lupus Erythematosus, and Patient With Cutaneous Lupus Erythematosus
Brief Title: A Study of KK4277 in Healthy Volunteers and Patients With Systemic Lupus Erythematosus and Cutaneous Lupus Erythematosus
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4277-001
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers; Systemic Lupus Erythematosus (SLE); Cutaneous Lupus Erythematosus (CLE)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Outcomes Assessor: pharmacokinetic person, pharmacodynamic analysis person and investigational drug administration person are unblinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KK4277 (Experimental)
  Interventions: Drug: KK4277

INTERVENTIONS:
Drug: Placebo — Placebo is administered single dose or multiple dose by IV or SC injection
  Arms: Placebo
Drug: KK4277 — KK4277 is administered single dose or multiple dose by IV or SC injection
  Arms: KK4277

SUMMARY:
Part 1 : To evaluate the safety and tolerability of a single intravenous (IV) or subcutaneous (SC) dose of KK4277 in healthy Japanese or non-Asian adult males.

Part 2 : To evaluate the safety and tolerability of repeated IV or SC administration of KK4277 in patients with Systemic lupus erythematosus (SLE) or Cutaneous lupus erythematosus (CLE).

ELIGIBILITY:
Inclusion Criteria: Part 1

* Voluntary written informed consent to participate in the study
* Japanese or non-Asian healthy men 18 to < 50 years at the time of informed consent
* BMI 18.5 to < 30.0 at screening

Inclusion Criteria: Part 2

* Voluntary written informed consent to participate in the study
* Age 18 years to < 75 years at the time of informed consent
* Weight over 40 kg and BMI 18.5 to < 35.0 at screening
* Patients who meet any of the following criteria

  1. Patients who meet the EULAR/ACR 2019 SLE classification criteria and have a diagnosis of SLE by screening
  2. Patients with CLE diagnosed by skin biopsy

Exclusion Criteria: Part 1

* Current illness requiring treatment
* History of or current respiratory disease, heart disease, gastrointestinal disease, kidney disease, liver disease, psychiatric disease, autoimmune disease, or Cancer.
* History or of current drug allergy

Exclusion Criteria:Part2

* Complications of active lupus nephritis(urinary column (granular column or red blood cell column), hematuria (>5 red blood cells/high power field, excluding other causes such as stones or infection), proteinuria >0.5 g/24 h, pyuria (>5 white blood cells/high power field excluding infection)) or active central nervous lupus (delirium, psychiatric symptoms, seizures, etc.)
* Patients with serious complications that are judged by the investigator or sub-investigator to affect the conduct and evaluation of the study.
* Patients with bacterial, viral, fungal, or parasitic infections recognized within 28 days prior to obtaining consent
* Patients with an infectious disease requiring hospitalization or IV administration of antimicrobial, antiviral, antifungal, or antiparasitic drugs within 24 weeks prior to obtaining consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Part 1 : from Day 1 through at most Day 113, Part 2: from Day 1 through at most Day 169
  For adverse events that occurred after administration of the investigational drug, number of subjects with AEs and occurrence frequency are evaluated.

SECONDARY OUTCOMES:
Profile of pharmacokinetics of serum KK4277 concentration | Part 1 : Day 1 (pre-dose, 0, 1, 6 hours after the start of administration), 2, 3, 4, 5, 6, 8, 15, 22, 29, 43, 57, 71, 85, 99, 113, Part 2 :Enrollment, Day1, 8, 15, 29, 43, 57, 71, 85, 99, 113, 141, 169
Time to the maximum concentration | Part 1 : Day 1 to Day 113, Part 2 : Day 1 to Day 169
The maximum concentration | Part 1 : Day 1 to Day 113, Part 2 : Day 1 to Day 169
Area under the concentration-time curve | Part 1 : Day 1 to Day 113, Part 2 : Day 1 to Day 169

CONTACTS AND LOCATIONS:
Overall Officials: Jun Kinoshita, Study Chair — Kyowa Kirin Co., Ltd.
Locations (23):
- Japan (21):
  - Fujita Health University Hospital, Kutsukake, Aichi-ken
  - Japan Community Health care Organization Chukyo Hospital, Minami, Aichi-ken
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Kyusyu University Hospital, Higashi, Fukuoka
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center, Minami, Kanagawa
  - Kitasato University Hospital, Minami, Kanagawa
  - National University Corporation Tohoku University Tohoku University Hospital, Aoba, Miyagi
  - Niigata University Medical & Dental Hospital, Chuo Ku, Niigata
  - University of the Ryukyus Hospital, Ginowan, Okinawa
  - Saitama Medical University Hospital, Moriyama, Saitama
  - Institute of Science Tokyo Hospital, Bunkyō-Ku, Tokyo
  - St. Luke's International Hospital, Chuo Ku, Tokyo
  - Showa Medical University East Hospital, Shinagawa-Ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Japan Institute for Health Security National Center for Global Health and Medicine, Shinjuku-Ku, Tokyo
  - Medical Co. LTA Sumida Hospital, Sumida-ku, Tokyo
  - Fukushima Medical University Hospital, Fukushima
  - Nagasaki University Hospital, Nagasaki
  - Juntendo University Nerima Hospital, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- South Korea (2):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.